CLINICAL TRIAL: NCT03471338
Title: Neuropsychological Management of Multiple Sclerosis: Benefits of a Computerised Semi-autonomous At-home Cognitive Rehabilitation Programme
Acronym: SEPIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2017-A01736-47
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
Keywords: multiple sclerosis; cognition; neuropsychology; cognitive rehabilitation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Patients benefit cognitive rehabilitation
  Interventions: Behavioral: Cognitive rehabilitation
- Standard Psychological care (Sham Comparator): Patients do not benefit cognitive rehabilitation
  Interventions: Behavioral: Standard Psychological care

INTERVENTIONS:
Behavioral: Cognitive rehabilitation — At-site inclusion visit: assessment of patient's eligibility by cognitive complaint questionnaire and BCcogSEP, VAPS and multiple errands test conducted by neuropsychologist.
  At-site baseline visit: assessment of quality of life (MUSIQOL), self-esteem (SEI), depression (MADRS), anxiety (HAMA), BICAMS: SDMT, CVLT-II, BVMTR, metacognition (MCQ-30), fatigue (EMIF-SEP), subjective sleep quality (PSQI) conducted by a neuropsychologist.
  At-home neuropsychological management (9 weeks): The patient performs the program (PRESCO software) on his computer autonomously at home at a rate of 3 sessions per week. A neuropsychologist performs at-home visits and weekly phone meetings to train the patient to the software, to encourage him to do exercises and to answer any software use-related questions.
  At-site follow-up visits: short and long-term retest of assessments performed in inclusion visit.
  Arms: Experimental Group
Behavioral: Standard Psychological care — At-site inclusion visit: assessment of patient's eligibility by cognitive complaint questionnaire and BCcogSEP, VAPS and multiple errands test conducted by neuropsychologist.
  At-site baseline visit: assessment of quality of life (MUSIQOL), self-esteem (SEI), depression (MADRS), anxiety (HAMA), BICAMS: SDMT, CVLT-II, BVMTR, metacognition (MCQ-30), fatigue (EMIF-SEP), subjective sleep quality (PSQI) conducted by a neuropsychologist.
  At-home neuropsychological management (9 weeks): A neuropsychologist performs at-home visits and weekly phone meetings consisting in discussion of the patient's cognitive disorders.
  At-site follow-up visits: short and long-term retest of assessments performed in inclusion visit.
  Arms: Standard Psychological care

SUMMARY:
Multiple sclerosis (MS) is a central nervous system inflammatory disease that causes a chronic and progressive physical handicap. Though primarily considered as a motor disease, it may, in 40 to 65% of cases, cause cognitive function deficits, concerning mainly attention, information processing speed, executive functions and memory. The impairment of these various functions may significantly impair the patients' social, professional and family lives. As such, the presence of cognitive difficulties is more frequently associated with the onset of anxio-depressive psychiatric symptoms and with reduced quality of life to the extent that it can be estimated via psychometric scales, or by a more qualitative approach. Recent research has focused, not on demonstrating the existence of cognitive disorders in MS, but rather on attempting to reduce their daily impact through cognitive rehabilitation programmes. While encouraging, the available results are relatively discordant and further work is required to demonstrate the actual efficacy of such programmes applied to daily life and of their long-term effects.

The main objective of this work is to evaluate, in patients suffering from MS and presenting with cognitive disorders and/or with complaints, the effect of an innovative computerised, semi-autonomous at-home cognitive rehabilitation programme, following care, on quality of life. The secondary objective is to estimate the improvement, or even stabilisation over time, of patients' cognitive performance and psycho-affective sphere.

In this randomised trial, the investigators plan to include 40 patients suffering from the RR and SP forms of MS, distributed to two groups paired by age, gender and socio-cultural level, one of which will benefit from computerised management, along with at-home support from a psychologist, while the other receives only the support.

This work is expected to provide two types of benefits. Firstly, to enable patients to better understand their cognitive function via daily management and as such to improve their quality of life and self-esteem. Secondly, to eventually allow more appropriate patient management by combining the quasi-systematic use of this programme with follow-up consultations with referring practitioners (neurologists, psychologists, etc.).

ELIGIBILITY:
Inclusion Criteria:

* MS defined according to the McDonald criteria revised in 2010
* Men and women aged between 18 and 65 years
* RR and SP forms
* Duration of progression ≤ 25 years
* EDSS ≤ 5.5
* Lack of disease activity as defined by the new Lublin criteria (2013)
* Cognitive complaint and/or cognitive disorders according to the investigator's judgement
* Impaired cognitive performance at least 1.65 SD below normative data at one test of the BCcogSEP battery
* French native language
* Owner of a laptop computer with Internet access
* Signing of the informed consent

Exclusion Criteria:

* - Other neurological, psychiatric or developmental diseases prior to the MS diagnosis
* Cranial trauma sequelae
* Chronic alcohol and/or drug consumption
* EDSS > 6
* Relapse and/or treatment with corticosteroids within the past month
* Persons deprived of liberty, minors, adults under wardship
* Cognitive examination within the past 6 months (including in particular all or some of the tests proposed by this project)
* Presence of dementia according to DSM V criteria, or of cognitive disorders preventing the patient from undergoing cognitive tests or performing cognitive rehabilitation exercises
* Any visual or motor deficit preventing the patient from undergoing cognitive tests or performing cognitive rehabilitation exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of cognitive rehabilitation on quality of life at short term. | 10 weeks
  Quality of life will be assessed by measuring the change of the scores of MUSIQOL (MUltiple Sclerosis International Quality Of Life) questionnaire between baseline and short-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on quality of life at long term. | 34 weeks
  Quality of life will be assessed by measuring the change of the scores of MUSIQOL (MUltiple Sclerosis International Quality Of Life) questionnaire between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.

SECONDARY OUTCOMES:
Efficacy of cognitive rehabilitation on self-esteem at short term. | 10 weeks
  Self-esteem will be assessed by measuring the change of the scores of the SEI (Self Esteem Inventory) scale between baseline and short-term. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on self-esteem long term. | 34 weeks
  Self-esteem will be assessed by measuring the change of the scores of the SEI (Self Esteem Inventory) scale between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on depression at short term. | 10 weeks
  Depression will be assessed by measuring the change of the scores of MADRS (Montgomery and Asberg Depression Rating Scale) questionnaire between baseline and short-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on depression at long term. | 34 weeks
  Depression will be assessed by measuring the change of the scores of MADRS (Montgomery and Asberg Depression Rating Scale) questionnaire between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on cognition at short term. | 10 weeks
  Cognition will be assessed by measuring the change of the scores of the BICAMS (Brief International Assessment for Multiple Sclerosis) battery between baseline and short-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on cognition at long term. | 34 weeks
  Cognition will be assessed by measuring the change of the scores of the BICAMS (Brief International Assessment for Multiple Sclerosis) battery between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on metacognition at short term. | 10 weeks
  Metacognition will be assessed by measuring the change of the scores of the MCQ-30 (Metacognitions Questionnaire-30) scale between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on metacognition at long term. | 34 weeks
  Metacognition will be assessed by measuring the change of the scores of the MCQ-30 (Metacognitions Questionnaire-30) scale between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on fatigue at short term | 10 weeks
  Fatigue will be assessed by measuring the change of the scores of the EMIF-SEP (Echelle Modifiée d'Impact de la Fatigue dans la Sclérose En Plaques) scale between baseline and short-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on fatigue at long term | 34 weeks
  Fatigue will be assessed by measuring the change of the scores of the EMIF-SEP (Echelle Modifiée d'Impact de la Fatigue dans la Sclérose En Plaques) scale between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on sleep at short term | 10 weeks
  Sleep will be assessed by measuring the change of the scores of the PSQI (Pittsburgh Sleep Quality Index) questionnaire between baseline and short-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on sleep at long term | 34 weeks
  Sleep will be assessed by measuring the change of the scores of the PSQI (Pittsburgh Sleep Quality Index) questionnaire between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on anxiety at short term. | 10 weeks
  Anxiety will be assessed by measuring the change of the scores of HAMA (HAMilton Anxiety) scale between baseline and short-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.
Efficacy of cognitive rehabilitation on anxiety at long term. | 34 weeks
  Anxiety will be assessed by measuring the change of the scores of HAMA (HAMilton Anxiety) scale between baseline and long-term visits. Efficacy will be assessed by comparing theses scores between groups A and B.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Defer, Pr, Principal Investigator — Neurology Department, Caen University Hospital
Locations (1):
- University Hospital of Caen, Caen, Calvados, France